CLINICAL TRIAL: NCT07138326
Title: Beeinflussung Der Resorption Von Arzneimitteln Bei Stoma Patient*Innen
Brief Title: Impact on the Absorption of Drugs in Ostomy Patients
Acronym: STAR
Status: Recruiting | Type: Observational
Sponsor: WiGeV Klinik Ottakring (Other)
Responsible Party: Sponsor
Other Study IDs: EK25008
Record Dates: First submitted 2025-06-20; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stoma Ileostomy; Ileostomy - Stoma; Colostomy - Stoma; Absorption; Pharmakokinetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Monitoring — Monitoring

SUMMARY:
Peroral administration is the preferred way of taking medication. However, the special absorption conditions in ostomy patients are generally not addressed in approval studies and there is also little other literature on this topic. These are usually case reports or studies on individual patients or very small patient collectives.

For medications with measurable clinical parameters, e.g. blood pressure, blood sugar, etc: Blood pressure, blood sugar, etc., these can be used to draw conclusions about any absorption problems. For medications without the possibility of a direct and objective assessment, the assessment is difficult due to the very low level of evidence. Drug groups without a direct physiological measure are e.g: Psy-chotropic drugs (antipsychotics, antidepressants, anxiolytics) and also the novel oral anticoagulants (NOACs).

The clinical trial´s results will answer the following questions:

* Are therapeutic blood levels of psychotropic drugs and NOACs achieved in ostomy patients when taken orally in the usual way?
* Are there differences between the measured levels of ileostomy and colostomy patients? Colostomy and ileostomy patients undergoing inpatient or outpatient treatment at the Klinik Ottakring are ready for inclusion. The blood samples will be obtained during medically indicated and performed blood draws within the scope of medical practice, so that no study-associated risks arise here.

Recorded and evaluated:

* Relevant patient data
* Plasma levels of the drugs under investigation in ostomy patients. The therapeutic range specified in the respective approval studies serves as the reference value. The results obtained are documented, evaluated and interpreted in an appropriate manner.

ELIGIBILITY:
Planned inclusion criteria:

* Male and female patients aged ≥18 years
* Belonging to a collective
* Ileostomy since ≥7d
* Colostomy since ≥7d The stoma must have been inserted at least 7d ago to ensure that a steady state concentration is achieved.
* Taking ≥1 of the following active substances since ≥7d:

  * Psychotropic drugs: citalopram, clozapine, duloxetine, escitalopram, melperone, mianserin, milnacipran, mirtazapine, olanzapine, paliperidone, paroxetine, pregabalin, prothipendyl, quetiapine, risperidone, sertraline, trazodone, venlafaxine
  * NOACs: edoxaban, rivaroxban, apixaban

Exclusion Criteria:

Insurmountable language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ileostomy and colostomy patients undergoing inpatient/outpatient treatment at Klinik Ottakring
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Achieved therapeutic serum levels in ostomy patients compared with the therapeutic ranges of the respective pivotal study | 18 month
  During a routine blood draw, an additional 2ml (Psychotropic drugs: citalopram, clozapine, duloxetine, escitalopram, melperone, mianserin, milnacipran, mirtazapine, olanzapine, paliperidone, paroxetine, pregabalin, prothipendyl, quetiapine, risperidone, sertraline, trazodone, venlafaxine)or 3.5 ml (NOACs: edoxaban, rivaroxban, apixaban)of blood is taken. In this sample, the drug levels are determined using a validated method ( LC-MS/MS (Psychotropic drugs) or chromogenic test (NOACs)). The drug level [µg/ml] determined in this way is compared with the therapeutic target range specified in the respective approval studies.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gläser, Dr, Study Chair — WiGeV Klinik Ottakring
Locations (1):
- WiGeV Klinik Ottakring, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No